CLINICAL TRIAL: NCT03921281
Title: Scalp Acupuncture Treatment for Motor Dysfunction in Children With Cerebral Palsy: Study Protocol for a Randomized Controlled Trial
Brief Title: Evaluating the Therapeutic Effect of Scalp Acupuncture Treatment for Motor Dysfunction in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHFudanU-1
Record Dates: First submitted 2019-04-13; First posted 2019-04-19 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Palsy; Motor Dysfunction; Acupuncture
Keywords: Cerebral palsy; Motor dysfunction; Scalp acupuncture treatment; Safety/Efficacy assessment
MeSH Terms: conditions — Cerebral Palsy; Neurologic Manifestations | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): The treatment group (n=38) will receive scalp acupuncture combined with rehabilitation treatment for 3 times per week for 12 weeks.
  Interventions: Other: scalp acupuncture treatment; Other: Rehabilitation Treatment
- control group (Other): The control group (n=38) will receive rehabilitation treatment for 3 times per week for 12 weeks.
  Interventions: Other: Rehabilitation Treatment

INTERVENTIONS:
Other: scalp acupuncture treatment — The parameters for scalp acupuncture are set as follows:
  1. Scalp acupoint selection: The Motor Area of Jiao's Scalp acupuncture and Si shencong (EX-HN1).
  2. Acupuncture manipulation: Disposable stainless steel needles will be manually inserted in at an approximately 15-degree angle to a depth of 1.5-2.0 cm respectively along the upper point and middle point of the motor area on the scalp. The acupuncture direction of Si shencong (EX-HN1) acupoint is toward the Baihui (GV20) acupoint. the needles will be rotated for at least 200 revolutions per minute for 1 minute every 20 minutes for a total of 60 minutes.
  3. Treatment course: three times a week, 12 weeks in total.
  Arms: treatment group
Other: Rehabilitation Treatment — The children with CP will receive the conventional rehabilitation programs as mentioned above. The rehabilitation programs will be carried out three times a week (once every other day) for 12 weeks, and every time, the rehabilitation treatment (PT and OT) will last approximately for 1 hour. All rehabilitation treatments will be carried out by qualified therapists.

SUMMARY:
The investigators design a Multi-center randomized, control study to evaluate the therapeutic effect of the scalp acupuncture treatment for motor dysfunction in children with cerebral palsy by using the following outcomes: motor function, activity of daily living, quality of life.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a well-recognized neurodevelopmental condition beginning in early childhood and persisting throughout the lifetime. Motor disorders are often accompanied by disturbances of sensation, cognition, communication, perception, behavior, and seizures The activities of daily living and social participation are limited in children with CP due to motor dysfunction, this greatly influences the CP patient's quality of life, and return to society.

Western conventional treatment of CP is multi-professional rehabilitation. In China, CP rehabilitation mainly develops the clinical mode of combining traditional Chinese medicine and western medicine. Acupuncture use as a complementary or alternative therapy has increased worldwide and has become widely applied to CP rehabilitation, which confirms that the efficacy of acupuncture can have a great impact on CP management. Many studies have shown that scalp acupuncture has a remarkable treatment efficacy on motor dysfunction in children with CP in China. But, Although acupuncture as a treatment for cp has become widely accepted and showed better clinical curative effect than conventional treatments, a Meta-Analysis published in 2018 based on clinical randomized controlled trials summarized that the clinical curative effect of acupuncture treatment in children with CP remains uncertain due to the small number of randomized controlled trials available and the small sample sizes. More high-quality and large-scale studies are still needed. The purpose of this study is to observe the therapeutic effect of scalp acupuncture treatment for motor dysfunction in children with CP by using the international general evaluation scales.

In this 12-week, assessor-blind, randomized, controlled study of scalp acupuncture as additional treatment with the rehabilitation treatment, a total of 76 children with cerebral palsy will be recruited. The patients will be randomly assigned to two different groups: 1) the treatment group and 2) the control group. The treatment group (n=38) will receive scalp acupuncture combined with rehabilitation treatment for 3 times per week for 12 weeks, and the control group (n=38) will receive rehabilitation treatment for 3 times per week for 12 weeks. Both groups will be evaluated at baseline, week4 (treatment 12), week 8 (treatment 24), week12(treatment 36) and week 24(follow-up) using GMFM scale, FMFM scale, PEDI scale and CP-QOL scale. The study will be conducted at Children's Hospital of Fudan University.

ELIGIBILITY:
Inclusion Criteria:

1. cerebral palsy patients between 12 and 72 months old
2. cerebral palsy was diagnosed according to the criteria of CP in international guidelines
3. children with CP of the spastic type
4. voluntary participation and informed consent signed

Exclusion Criteria:

1. visual, auditory and mental disorders, affecting the rehabilitation assessment
2. the child with epilepsy who is not under control with medication
3. bleeding tendencies
4. being oversensitive to acupuncture
5. use of muscle relaxants or herbal therapies during the study period
6. participation in another clinical trial

Ages: 12 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline GMFM at 4 weeks, 8 weeks and 12 weeks | The GMFM will be assessed at baseline, interventions period (4 weeks, 8 weeks and 12 weeks) and fellow-up period at (24 weeks).
  The Gross Motor Function Measure (GMFM) is a standardized observational instrument designed to assess the gross motor function of children with CP. It is divided into five sections: Lying and Rolling, Sitting, Crawling and Kneeling, Standing, and Walking, Running and Jumping. Each item is on the basis of four levels: 0=does not initiate, 1=initiates, 2=partially completes, 3=completes or NT=not tested. The total score is a summation of the scores in the five areas by the Gross Motor Ability Estimator software (GMAE Version 1.0.)
Change from Baseline FMFM at 4 weeks, 8 weeks and 12 weeks | The FMFM will be assessed at baseline, interventions period (4 weeks, 8 weeks and 12 weeks) and fellow-up period at (24 weeks).
  The Fine Motor Function Measure (FMFM) assessment scale is used to evaluate the fine motor activities of children with CP, including the upper limb activities and sensory ability. This scale includes five domains, namely audiovisual tracking ability(5 items), upper limb joint's ability(9 items), grasping ability(10 items), operation ability(13 items)and hand-eye coordination(24 items). Each item is on the basis of four levels: 0=does not initiate, 1=initiates, 2=partially completes, 3=completes. The total score(0～100 points) is a summation of the scores in the five areas.

SECONDARY OUTCOMES:
Change from Baseline PEDI at 4 weeks, 8 weeks and 12 weeks | PEDI will be assessed at baseline, interventions period (4 weeks, 8 weeks and 12 weeks) and fellow-up period at (24 weeks).
  Pediatric Evaluation of Disability Inventory (PEDI) measures both functional performance and capability within three domains of (1) self-care, (2) mobility, and (3) social function in two categories, that is, the Functional Skills Scale (FSS), Caregiver Assistance Scale (CAS), and Modifications Scale. FSS covers 40 diverse content areas assessed using 197 items scored unable (0) or capable (1). The self-care domain comprises 73 items. The mobility domain has 59 items. The social function domain has 65 items. CAS It covers 20 diverse content areas assessed using 20 items scored on the following escalating 6-point scale: independent, supervision, minimal help, moderate help, maximum help, and total help. The items cover the self-care domain (n = 8), mobility domain (n = 7), and social function domain (n = 5). Modifications Scale measures any environmental or technical modifications needed to enhance the child's function.
Change from Baseline CPQOL at 4 weeks, 8 weeks and 12 weeks | CPQOL will be assessed at baseline, interventions period (4 weeks, 8 weeks and 12 weeks) and fellow-up period at (24 weeks).
  The cerebral palsy quality of life questionnaire for children contains 66 items in seven domains: Social well-being and acceptance (SWB), Functioning (FUN), Participation and physical health (PART), Emotional well-being (EWB), Access to services (ACCESS), Pain and feeling about disability (PAIN), and Family health (FAMILY). Almost all of the items have the following item stem: 'How do you think your child feels about. . .' and a 9-point rating scale, where 1 = very unhappy, 3 = unhappy, 5 = neither happy nor unhappy, 7 = happy, and 9 = very happy.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, Ph.D., Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Because our data is managed by the clinical trial unit. We will respect the opinions of the clinical research unit management committee and the subjects, which will ultimately decide whether to share the study data with other researchers.

REFERENCES:
- [Derived] Wang J, Shi W, Khiati D, Shi B, Shi X, Luo D, Wang Y, Deng R, Huang H, Li J, Yan W, Yang H. Acupuncture treatment on the motor area of the scalp for motor dysfunction in children with cerebral palsy: study protocol for a multicenter randomized controlled trial. Trials. 2020 Jan 6;21(1):29. doi: 10.1186/s13063-019-3986-z. PMID 31907027